CLINICAL TRIAL: NCT07228676
Title: INSPIRatory Efforts Estimation Under High-flow Nasal Oxygen: a Pilot Study
Brief Title: INSPIRatory Efforts Estimation Under High-flow Nasal Oxygen
Acronym: INSPIRE-Pilot
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-A01663-46
Record Dates: First submitted 2025-09-17; First posted 2025-11-14 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Oxygen; Respiratory Insufficiency; Work of Breathing; Dyspnea
Keywords: high-flow nasal oxygen; respiratory failure; inspiratory efforts; dyspnea
MeSH Terms: conditions — Respiratory Insufficiency; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Critically ill patients treated with HFNO (Experimental): Patients treated with HFNO for less than 24 hours in ICU
  Interventions: Other: Non-invasive estimation of inspiratory effort

INTERVENTIONS:
Other: Non-invasive estimation of inspiratory effort — As soon as possible after inclusion and 2 hours later, tracings of pressure and flow delivered by the HFNO device will be collected using a noninvasive extracorporeal sensor placed between the nasal cannulas and the HFNO device, as well as vital signs and dyspnea. At each visit, tracings will be collected for 10 minutes using the HFNO flow set by the clinician and for 10 minutes using an HFNO flow of 30 L/min allowing the patient breathing mouth closed. During the recordings, patients will be monitored closely at the bedside by the investigator. Estimated inspiratory efforts under HFNO will be calculated a posteriori. HFNO failure (intubation or reintubation) will be assessed at day 7 of inclusion. Vital status will be assessed at day 28 of inclusion.

SUMMARY:
High-flow nasal oxygen (HFNO) is recommended as first-line treatment to prevent intubation in acute hypoxemic respiratory failure and to prevent reintubation after extubation. Accumulating data suggest that strong inspiratory efforts and their persistence are associated with HFNO failure. However, tools to monitor continuously and noninvasively inspiratory efforts are lacking. The investigators have developed an algorithm estimating noninvasively inspiratory efforts under HFNO. This pilot study aims at testing the feasibility of estimating inspiratory efforts in patients treated with HNFO.

DETAILED DESCRIPTION:
High-flow nasal oxygen (HFNO) is recommended as first-line treatment to prevent intubation in acute hypoxemic respiratory failure and to prevent reintubation after extubation (alone in patients at low-risk of extubation failure, alternating with noninvasive ventilation in patients at high-risk of extubation failure). It consists in delivering high flow of heated and humidified gas enriched with oxygen through nasal cannulas. However, HFNO failure occurs in 30 to 50% of cases in acute hypoxemic respiratory failure and 10 to 20% of cases after extubation.

Accumulating data suggest that strong inspiratory efforts and their persistence are associated with HFNO failure. However, the monitoring of inspiratory efforts is challenging, especially in patients breathing spontaneously through the nose under HFNO. On a bench study, the investigators have developed an algorithm estimating noninvasively inspiratory efforts under HFNO based on the analysis of tracings of pressure and flow delivered by the HFNO device using an extracorporeal sensor. The coefficient of determination of the algorithm was high (R2=0.92). This pilot study aims at testing the feasibility of estimating inspiratory efforts in patients treated with HNFO.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 yo admitted to the intensive care unit
* Treated with HFNO for less than 24h to prevent intubation of reintubation
* Affiliated to social insurance
* Consent to participate in the study

Exclusion Criteria:

* Do-not-intubate order at inclusion
* Already included in the study
* Under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-29 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The detection of estimated inspiratory efforts under HFNO in patients breathing through the nose at a flow rate of 30 L/min in at least 16 of the 20 (≥ 80%) patients included. | Day 1
  Inspiratory efforts will be calculated a posteriori using the algorithm developed on the bench, based on the pressure and flow signals delivered by the HFNO device collected during the first recording.

SECONDARY OUTCOMES:
Inspiratory efforts estimated under HFNO in patients breathing through the nose at a flow rate of 30 L/min between HFNO success and failure in the overall population and in each subgroup (prevention of intubation and of reintubation) | Day 7
  Inspiratory efforts estimated under HFNO in patients breathing through the nose at a flow rate of 30 L/min will be calculated a posteriori using the algorithm developed on the bench based on the pressure and flow signals delivered by the HFNO device collected during the first recording.
  HFNO failure is defined as intubation or reintubation or death at day 7 after inclusion.
Inspiratory efforts estimated under HFNO in patients breathing through the nose at a flow rate of 30 L/min between survivors and non survivors at day 28 in the overall population and in each subgroup (prevention of intubation and of reintubation) | Day 28
  Inspiratory efforts estimated under HFNO in patients breathing through the nose at a flow rate of 30 L/min will be calculated a posteriori using the algorithm developed on the bench, based on the pressure and flow signals delivered by the HFNO device collected during the first recording.
The change in inspiratory efforts between the 2 visits between HFNO success and failure in the overall population and in each subgroup (prevention of intubation and of reintubation) | Day 7
  The change in inspiratory efforts is defined as the decrease in estimated inspiratory efforts under HFNO in patients breathing through the nose at a flow rate of 30 L/min calculated a posteriori using the algorithm developed on the bench based on the pressure and flow signals delivered by the HFNO device between the first and second recording.
  HFNO failure is defined as intubation or reintubation or death at day 7 after inclusion.
The change in inspiratory efforts between the 2 visits between survivors and non survivors at day 28 in the overall population and in each subgroup (prevention of intubation and of reintubation) | Day 28
  The change in inspiratory efforts is defined as the decrease in estimated inspiratory efforts under HFNO in patients breathing through the nose at a flow rate of 30 L/min calculated a posteriori using the algorithm developed on the bench based on the pressure and flow signals delivered by the HFNO device between the first and second recording.
Inspiratory efforts estimated under HFNO according to dyspnea at each visit | Day 1
  Inspiratory effort estimated under HFNO in patients breathing through the nose at a flow rate of 30 L/min at each recording, and dyspnea score.
  Dyspnea is defined as a value ≥ 4/10 on a numerical rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Céline ABONNEAU, Study Chair — Poitiers University Hospital
Locations (1):
- Poitiers University Hospital, Poitiers, France

IPD SHARING:
Plan to Share IPD: No
This pilot study will be followed by a larger prospective observational study.